CLINICAL TRIAL: NCT01112293
Title: A Phase II Trial of Anti-TGF Monoclonal Antibody (GC1008) in Relapsed Malignant Pleural Mesothelioma (MPM))
Brief Title: Anti-TGF Monoclonal Antibody (GC1008) in Relapsed Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03510
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Pleural Malignant Mesothelioma
Keywords: Subjects who have pleural malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational drug infusion-for safety and effectiveness (Experimental): Phase II, Single-Arm, Multi-Site study. All subjects will receive the investigational agent, GC1008 in 3 week cycles of treatment
  Interventions: Drug: GC1008

INTERVENTIONS:
Drug: GC1008 — GC1008 is a human IgG4 kappa monoclonal antibody capable of neutralizing all mammalian isoforms of TGFbeta (i.e., beta1, beta 2 and beta 3). GC1008 is a high affinity antibody with dissociation constants (Kds) of 1.8 nM, 2.8 nM and 1.4 nM for TGF1,2,and 3, respectively.
  Other Names: IgG4 kappa monoclonal antibody

SUMMARY:
This study is being conducted to evaluate the overall safety and effectiveness of an investigational drug, GC1008, in patients with mesothelioma. An investigational drug is one that has not been approved by the FDA. Approximately 40 people will be enrolled on this study at the University of Pennsylvania (Main Institution/Coordinating Site) and the University of Chicago (Participating Institution). We expect about 20 subjects to be enrolled at each institution.

DETAILED DESCRIPTION:
Primary: - To assess progression-free survival rate at three months.

Secondary: - To determine the toxicity and safety of systemic infusion of anti-TGF beta antibody at three-week dosing intervals. - To assess time to progression and overall survival - to assess response rate using Modified RECIST Criteria for Mesothelioma Additional Objectives: - To assess efficacy using serial measurements of serum [and intrapleural, if indwelling catheter in place] biomarkers, including serum-mesothelin related peptide (SMRP/Mesomark®) and osteopontin. - To assess systemic [and intrapleural if indwelling catheter in place] humoral anti-tumor immune responses after repeated anti-TGF beta antibody instillation. - To assess systemic [and intrapleural, if indwelling catheter in place] TGF beta, and other cytokine levels after repeated anti-TGF beta antibody instillation. - To assess biologic response measurements of TGF beta blockade from serum tests and from pleural fluid or biopsy tissue if this is available.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically [histologically or cytologically] documented pleural malignant mesothelioma.

Patients must have had at least one, but no more than two prior systemic therapies, at least one of which contained pemetrexed.

* Documented progressive disease evaluable by Modified RECIST criteria. [Progressive symptoms after 1st line therapy in the absence of objective progression are acceptable as a criterion for enrollment]. Patients who have had previous extrapleural pneumonectomy and disease recurrence will be eligible if they have no other exclusion criteria.
* ECOG Performance status of 0 or 1.
* Greater or equal to 18 years of age.
* Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial.
* Must be able and willing to give written informed consent. Patients may not be consented by a durable power of attorney.
* Serum albumin greater or equal to 2.5
* Adequate organ function
* Patients must have negative tests for human immunodeficiency virus (HIV) and for hepatitis viruses B and C (antibody and/or antigen) unless the result is consistent with prior vaccination or prior infection with full recovery.
* At the time of enrollment, patients must be greater than 3 weeks since major surgery, radiotherapy, chemotherapy (greater or equal to 6 weeks if they were treated with a nitrosourea, mitomycin or monoclonal antibody), immunotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to less than or equal to Grade 1, exclusive of alopecia. Concurrent non-protocol cancer therapy is not permitted. (In patients who received long acting agents, a treatment free interval of 2 half lives should be considered.) Note: Although a patient can be entered by these criteria, if a patient is less than 3-6 months from radiotherapy or talc pleurodesis, FDG-PET scanning will not be useful. 12).

Exclusion Criteria:

* Known central nervous system (CNS) metastases, meningeal carcinomatosis, malignant seizures, or a disease that either causes or threatens neurologic compromise (e.g., unstable vertebral metastases).
* Presence of pericardial effusion
* Rapidly re-accumulating, symptomatic malignant pleural effusions status-post thoracentesis or pleural catheter insertion that requires immediate mechanical or chemical pleurodesis for adequate palliation.
* Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or use of anti-coagulation therapy (including lovenox, warfarin, or anti platelet agents such as aspirin [with the exception of low dose ASA ~ 81 mg/d] , clopidogrel, ticlopidine, dipyridamole, and other agents used to induce long-acting platelet dysfunction). Patients with a history of deep venous thrombosis may participate if successfully treated, completely resolved, and no treatment has been given for greater than 4 months.
* Pregnant or nursing women, due to the unknown effects of GC1008 on the developing fetus or newborn infant.
* Other active invasive malignancy requiring ongoing therapy.
* Patients with an organ transplant, including those that have received an allogeneic bone marrow transplant.
* Use of investigational agents within 4 weeks prior to study enrollment (within 6 weeks if the treatment was with a long-acting agent such as a monoclonal antibody).
* Patients on immunosuppressive therapy
* Significant or uncontrolled medical illness, such as congestive heart failure (CHF), myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction.

Patients with a remote history of asthma or active mild asthma may participate.

* Active infection, including active herpes zoster, as well as unexplained fever (temperature 38.1C), or antibiotic therapy within 1 week prior to enrollment.
* Systemic autoimmune disease (e.g., systemic lupus erythematosus, active rheumatoid arthritis, etc.).
* Positive stool fecal occult blood test (patients who are positive will need a standard GI work-up consisting of an Esophagogastroduodenoscopy (EGD) and Colonoscopy) prior to enrollment to rule out possible reasons for bleeding. A patient will be eligible with negative results for both exams.
* Active GI bleeding within past 5 years other than due to benign anorectal causes such as hemorrhoids, fissures and stricture.
* A known allergy to any component of GC1008.
* Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Stevenson, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: 3-month Progression Free Survival Rate
Description: The fraction of subjects surviving 3 months without disease progression.
Time Frame: 3 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants | 3

2. Secondary Outcome: Toxicity and Safety of Systemic Infusion of Anti-TGF Antibody
Description: The toxicity and safety of systemic infusion of anti-TGF antibody at three-week dosing intervals. Number subjects with Grade 2 and Grade 3/4 treatment related toxicities.
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Number; unit: participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
participants
  Grade 2 Treatment Related Toxicities | 4
  Grade 3/4 Treatment Related Toxicities | 3

3. Other Pre Specified Outcome: Time to Progression and Overall Survival
Description: Assessment of time to disease progression and overall survival
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Months
  Time to Progression | 1.4 [1.2 to NA] — Data was reported as a one sided Confidence Interval, so there is no upper limit interval reported
  Overall Survival | 12 [7.17 to 14.43]

4. Other Pre Specified Outcome: Response Rate Using Modified RECIST Criteria for Mesothelioma
Description: Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in RECIST. The response assessment is based on the presence, absence, or unequivocal progression of the lesions.
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants | 0

5. Other Pre Specified Outcome: Number of Participants With a Change of Serum Biomarkers After Therapy
Description: Evaluation of changes after treatment therapy to a number of potential blood biomarkers of TGF-β effect (serum osteopontin, serum hyaluronan, serum MMP-1, serum MMP-7, serum IL-6, plasma CCL18, plasma VEGF, and plasma PAI-1). Animal models predict acute changes in TGF-β levels in blood associated with changes in serum biomarkers.
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants
  Change in serum osteopontin after treatment | 0
  Change in serum hyaluronan after treatment | 0
  Change in serum MMP-1 after treatment | 0
  Change in serum MMP-7 after treatment | 0
  Change in serum IL-6 V after treatment | 0
  Change in plasma CCL18 v after treatment | 0
  Change in plasma VEGF after treatment | 0
  Change in plasma PAI-1 after treatment | 0

6. Other Pre Specified Outcome: Number of Participants With Systemic Humoral Anti-tumor Immune Response After Repeated Anti-TGFβ Antibody Instillation
Description: Comparing antibody bands in pre-treatment versus post-treatment serum
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants | 6

7. Other Pre Specified Outcome: Assessment of Systemic TGFβ After Repeated Anti-TGFβ Antibody Installation
Description: The number of participants with significant change in percentage of circulating CD4+ T regulatory cells, marked by expression of FOXP3 after treatment. TGFβ has been implicated in the formation of T regulatory cells, and the blockade of TGFβ in animal models can inhibit the formation of T regulatory cells.
Time Frame: 18 months
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants | 0

8. Other Pre Specified Outcome: Biologic Response Measurements of TGFβ Blockade
Description: Number of participants who demonstrated upregulation of NK cell receptors 3 weeks after treatment. There are data that show anti-TGFβ antibodies can upregulate NK cell receptors in patients with chronic viral infections. TGFβ blockade was measured in samples of serum tests and from pleural fluid or biopsy if available.
Time Frame: 3 weeks
Population: Outcome analysis presented in manuscript of results of trial based on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of first administration of study product until 30 days of the last administration of study product, approximately 1 year and 5 months.
Arm/Group | Investigational Drug infusion-for Safety and Effectiveness
All-Cause Mortality (participants affected / at risk) | 12/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Drug infusion-for Safety and Effectiveness (N=14)
Nausea (Gastrointestinal disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (Cardiac disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Disease Progression (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (Blood and lymphatic system disorders) | 1 (1)
(General disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Drug infusion-for Safety and Effectiveness (N=14)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Fatigue (Cardiac disorders) | 9 (11)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back Pain (Injury, poisoning and procedural complications) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Mucosal Infection (Infections and infestations) | 1 (1)
(General disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Edema Limbs (General disorders) | 1 (1)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial include small sample size and lack of post-tumor treatment samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes